CLINICAL TRIAL: NCT06850064
Title: Efficacy and Safety of Pulsed Field Ablation in Refractory Bisththis-dependent Atrial Flutter: Pulsed Field Ablation Vs. Radiofrequency Ablation: a Preliminary Randomized Controlled Study
Brief Title: Efficacy and Safety of Pulsed Field Ablation in Refractory Mitral Isthmus-dependent Atrial Flutter: Pulsed Field Ablation Vs. Radiofrequency Ablation: a Preliminary Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIDAF-PFA vs RF
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Mitral Isthmus; PFA
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency ablation unit (Active Comparator): The patient underwent radiofrequency ablation treatment. After electrophysiological examination, radiofrequency ablation was performed.
  Interventions: Procedure: Radiofrequency ablation
- The pulse field ablation group (Experimental): The pulse field ablation group will undergo pulse field ablation of the mitral valve commissure.
  Interventions: Procedure: Pulse Field Ablation (PFA)

INTERVENTIONS:
Procedure: Pulse Field Ablation (PFA) — The pulse field ablation group will undergo pulse field ablation of the mitral valve commissure.
  Arms: The pulse field ablation group
Procedure: Radiofrequency ablation — In the radiofrequency ablation group, patients will undergo radiofrequency ablation targeted at the mitral valve commissure.
  Arms: Radiofrequency ablation unit

SUMMARY:
Efficacy and safety of pulsed field ablation in refractory mitral isthmus-dependent atrial flutter: pulsed field ablation vs. radiofrequency ablation: a preliminary randomized controlled study

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of pulse field ablation (PFA) versus radiofrequency ablation (RFCA) in improving mitral valve commissural block rate and atrial tachycardia recurrence rate in patients with refractory mitral valve commissural-dependent atrial flutter.

Study Design:

Randomized Groups: Patients will be randomly assigned to two groups:

Pulse Field Ablation (PFA) Group Radiofrequency Ablation (RFCA) Group

ELIGIBILITY:
Inclusion Criteria:

1.Patients aged ≥18 years. 2.Diagnosed with persistent symptomatic refractory mitral valve commissural-dependent atrial flutter. Refractory mitral valve commissural-dependent atrial tachycardia is defined as:

1. Failure of drug therapy: At least one Class I or III antiarrhythmic drug (e.g., propafenone, amiodarone) fails to effectively control or prevent episodes.
2. Failure of catheter ablation: At least one previous attempt at radiofrequency catheter ablation (RFCA) targeting the mitral valve commissure has been unsuccessful (either due to recurrence post-procedure or failure to achieve bidirectional block at the commissure).

3.Intolerant to at least one antiarrhythmic drug (AAD). 4.The patient must be capable of and willing to provide written informed consent to participate in this study.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Presence of left atrial thrombus on preoperative imaging.
3. Life expectancy less than 1 year.
4. Coagulation disorders or contraindications to anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Achieve persistent mitral isthmus block | Immediate post-operative mitral isthmus block rate.
  After mitral isthmus block, wait for 20 minutes, and obtain persistent MI block after the waiting period.

SECONDARY OUTCOMES:
Episodes of atrial fibrillation, atrial flutter, or atrial tachycardia lasting ≥30 seconds occurred. | During the 3-month post-operative follow-up.
  During the 3-month post-operative follow-up, episodes of atrial fibrillation, atrial flutter, or atrial tachycardia lasting ≥30 seconds occurred.
The safety endpoint | During the 3-month post-operative follow-up.
  The safety endpoint is a composite of major safety events, including pericardial tamponade or perforation, peripheral or organ thromboembolism, stroke or transient ischemic attack, persistent (lasting longer than hospitalization) phrenic nerve paralysis, atrioventricular block, pericarditis, vascular access complications requiring intervention, myocardial infarction, angina, myocardial infarction, coronary artery spasm, atrial-esophageal fistula, and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No